CLINICAL TRIAL: NCT01608074
Title: Radical Fimbriectomy for Young BRCA Mutation Carriers at Risk of Pelvic Serous Carcinoma
Brief Title: Radical Fimbriectomy for Young BRCA Mutation Carriers
Acronym: Fimbriectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: CTD-CNO (Unknown); Laboratoire PRISM (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FIMBRIECTOMIE-1106
Record Dates: First submitted 2012-05-15; First posted 2012-05-30 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation; Hereditary Breast and Ovarian Cancer
Keywords: BRCA1; BRCA2; Prophylactic surgery; Salpingectomy; Fimbriectomy
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRCA mutation carriers (Experimental): Women with BRCA1 or BRCA 2 mutation or a family history of breast/ovarian cancer.
  Radical fimbriectomy. Histopathology SEE-FIM
  Interventions: Procedure: Radical fimbriectomy; Other: Histopathology SEE-FIM

INTERVENTIONS:
Procedure: Radical fimbriectomy — Laparoscopic bilateral radical fimbriectomy :
  Complete resection of the tubes, from the uterine tube (up against the uterus) to the fimbriae, with resection of the part of the ovary adjacent to the ovarian fimbriae (adhering to the ovary)
Other: Histopathology SEE-FIM — Anatomopathological study of surgical specimens
  Other Names: Sectioning and Extensively Examining the FIMbria

SUMMARY:
Some BRCA-mutated women are reluctant to undergo laparoscopic bilateral salpingo-oophorectomy. The goal of the bilateral laparoscopic radical fimbriectomy the investigators suggest, is to suppress the tubal source of possible dysplastic cells from which can stem this high grade tumor, while preserving a natural ovarian hormonal secretion.

DETAILED DESCRIPTION:
Most of ovarian carcinomas related to BRCA 1 or 2 mutations are of fallopian tube origin and especially from its distant part called the fimbria. These tubal, ovarian or primary peritoneal carcinomas are quite always of high grade serous type. They cannot be effectively screened due to the quickness of their evolution. In this context, a laparoscopic bilateral salpingo-oophorectomy (BSO) is the recommended prophylactic procedure.

Some BRCA-mutated women are reluctant to undergo this procedure considering the numerous adverse effects on body and quality of life, especially when hormonal replacement is forbidden. This refusal makes them at risk of developing a serous pelvic carcinoma.

The goal of the bilateral laparoscopic radical fimbriectomy the investigators suggest, is to suppress the tubal source of possible dysplastic cells from which can stem this high grade tumor, while preserving a natural ovarian hormonal secretion

ELIGIBILITY:
Inclusion Criteria:

* Woman aged over 35 years
* When project of childbearing is fulfilled
* With a BRCA 1 or 2 mutation, or a family history of breast/ovarian cancer
* Unprepared to undergo bilateral annexectomy
* With or without breast cancer
* Patient affiliated to health insurance
* Dated and signed informed consent

Exclusion Criteria:

* Menopausal woman defined as :

Bilateral oophorectomy without hysterectomy and amenorrhea more than 12 months and/or FSH> 20 UI/l History of hysterectomy and FSH> 20 UI/l

* Pregnant or breastfeeding woman

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2033-08 (Estimated); Study Completion 2033-08 (Estimated)

PRIMARY OUTCOMES:
Rate of pelvic cancer | an expected average of 15 years
  Number of ovarian or primary serous peritoneal carcinoma occuring between fimbriectomy and menopause

SECONDARY OUTCOMES:
Morbidity associated with the radical prophylactic fimbriectomy | Up to 30 days after the surgery
  Morbidity will be assessed according to the Clavien-Dindo classification up to 30 days after the procedure and according to the NCI-CTCAE v4.0 grading scale beyond that time
Rate of occult lesions on fimbriectomy specimens and secondary oophorectomy specimens | Within 1 month after fimbriectomy, and within 1 month after oophorectomy
  Number of serous tubal intraepithelial carcinoma or invasive carcinomas on the operative specimens
Incidence of breast cancer on patients without breast cancer before fimbriectomy, and incidence (de novo or recurrence) of breast cancer on the overall study population | an expected average of 15 years
  Number of cases of breast cancer or breast cancer recurrence observed
Rate of secondary oophorectomies and associated morbidity, and reasons for oophorectomy if decided before the age of 50 et before menopausis | an expected average of 15 years
  Number of oophorectomies and time between fimbriectomy and oophorectomy Complications according to NCI-CTCAE v4.0 grading scale
Proteomic profile of tissues from radical fimbriectomy | Up to 7 years after sample collection
  Immunostaining is realised on sections of ovary portion, fimbriae and fallopian tubes, then tumoral zones are selected for spatially resolved gun microproteomic analysis
Proportion of menopausal women before oophorectomy or at the LPLV without oophorectomy, and rate patients who experienced early menopause (before the age of 40) | an expected average of 15 years
  Number of cases of menopausis an early menopausis observed
Proportion of benign histological abnormalities on radical Fimbriectomy specimens | Within 1 month after fimbriectomy
  Number of benign histological abnormalities on the operative specimens
Patient's satisfaction at distance from Radical Fimbriectomy | Up to 10 years
  Patient satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: Carlos MARTINEZ-GOMEZ, MD, Principal Investigator — Centre Oscar Lambret
Locations (14):
- France (14):
  - Polyclinique du Parc Rambot, Aix-en-Provence
  - Institut Bergonié, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - CHR-U, Lille
  - Clinique du Bois - Bourgogne Center, Lille
  - Hospices Civils de Lyon, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Centre Henri Becquerel, Rouen
  - IUCT-O Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif
  - Hôpital Privé VA, Villeneuve-d'Ascq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wisztorski M, Aboulouard S, Roussel L, Duhamel M, Saudemont P, Cardon T, Narducci F, Robin YM, Lemaire AS, Bertin D, Hajjaji N, Kobeissy F, Leblanc E, Fournier I, Salzet M. Fallopian tube lesions as potential precursors of early ovarian cancer: a comprehensive proteomic analysis. Cell Death Dis. 2023 Sep 30;14(9):644. doi: 10.1038/s41419-023-06165-5. PMID 37775701
- [Result] Leblanc E, Narducci F, Ferron G, Mailliez A, Charvolin JY, Houssein EH, Guyon F, Fourchotte V, Lambaudie E, Crouzet A, Fouche Y, Gouy S, Collinet P, Caquant F, Pomel C, Golfier F, Vaini-Cowen V, Fournier I, Salzet M, Tresch E, Probst A, Lemaire AS, Deley ML, Hudry D. Prophylactic Radical Fimbriectomy with Delayed Oophorectomy in Women with a High Risk of Developing an Ovarian Carcinoma: Results of a Prospective National Pilot Study. Cancers (Basel). 2023 Feb 10;15(4):1141. doi: 10.3390/cancers15041141. PMID 36831483